CLINICAL TRIAL: NCT06821126
Title: Randomized, Controlled, Multicenter Phase I/II Study Comparing the Safety and Immunogenicity of a Booster Dose of an Intranasal COVID-19 Vaccine Expressing SARS-CoV-2 N/S Recombinant Proteins With a Booster Dose of COVID-19 mRNA Vaccine in Healthy Adults (MUCOBOOST)
Brief Title: Study Comparing Safety and Immunogenicity of Intranasal COVID-19 Vaccine and mRNA Booster in Healthy Adults
Acronym: MUCOBOOST
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University Hospital, Tours (Cosponsor) (Unknown); UMS 54 MART (Unknown); INSERM CIC 1415 (Unknown); LovalTech (Unknown); INSERM U1259 MAVIVHe (Unknown); BioMAP - UMR ISP 1282 - Tours University - INRAE (Unknown); Virology unit, University Hospital, Tours (Unknown); I-REIVAC Innovative Clinical Research Network In Vaccinology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DR230330 - ANRS0514s MUCOBOOST; 2024-510589-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-28; First posted 2025-02-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: COVID-19; Healthy; Nasal; vaccine; intranasal
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase I : Dose escalation Phase II : open label, superiority, controlled, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVT-001 (Experimental): One booster dose of the intranasal vaccine LVT-001 administered as a nasal spray in each nostril at Day 0.
  Phase I - 3 cohortes with dose escalation (low, middle and high doses) Phase II - 1 arm at the selected dose
  Interventions: Biological: LVT-001
- Comirnaty (Active Comparator): One booster dose of the intramuscular COVID-19 mRNA vaccine (Pfizer-BioNTech - recommended at the beginning of the Phase II in France) at Day 0.
  Interventions: Biological: Cormirnaty

INTERVENTIONS:
Biological: LVT-001 — Intranasal administration
  Arms: LVT-001
Biological: Cormirnaty — Intramuscular administration
  Arms: Comirnaty

SUMMARY:
This Phase I/II trial in France evaluates safety and immunogenicity of a booster dose of an intranasal COVID-19 vaccine (LVT-001) versus a booster dose of a COVID-19 mRNA vaccine (Pfizer-BioNTech) in healthy adult volunteers.

As a first-in-human trial, Phase I will assess the safety and immunogenicity of three escalating doses of the LVT-001 vaccine across 3 cohorts of 12 volunteers per dose level.

Based on cumulative data collected up to Day 28 visit from the last included participant in the Phase I, the go/no-go decision for Phase II and selection of the optimal dose will be performed.

Phase II will then evaluate the immunogenicity of the selected intranasal dose of LVT-001 vaccine, compared to the standard of care of intramuscular COVID-19 mRNA Pfizer-BioNTech booster.

DETAILED DESCRIPTION:
This is a randomized, comparative, multicenter, open-label, phase I/II trial in France evaluating the safety and immunogenicity of a booster dose of an intranasal COVID-19 vaccine (LVt-001) versus a booster dose of a COVID-19 mRNA vaccine (Pfizer-BioNTech) in healthy adult volunteers.

Phase I dose escalating - Primary Objective: To evaluate the safety of three escalating doses of a boost of an intranasal COVID-19 vaccine (LVT-001) expressing SARS-CoV-2 N/S recombinant protein in healthy volunteers.

Phase II superiority trial - Primary Objective: To evaluate, using nasal swabs, the superiority of a booster dose of the selected intranasal COVID-19 vaccine (LVT-001) expressing SARS-COV-2 N/S recombinant protein versus a booster dose of the intramuscular COVID-19 mRNA vaccine (Pfizer-BioNTech) in healthy adult volunteers in term of mucosal humoral immune response at Day 28.

Trial population: A total of 36 and 202 healthy volunteers will be enrolled in Phase I and Phase II, respectively.

Interventions:

Phase I: The investigational medicinal product is the intranasal recombinant protein vaccine LVT-001 administered at Day 0 in each nostril:

* Cohort A (12 participants): 20 µg
* Cohort B (12 participants): 60 µg
* Cohort C (12 participants): 120 µg

Phase II: Two investigational medicinal products will be compared:

* The selected dose of the intranasal recombinant protein vaccine LVT-001, administered at Day 0 in each nostril.
* The intramuscular COVID-19 mRNA vaccine (Pfizer-BioNTech), administered as the standard of care booster.

Expected Outcomes and Safety Considerations:

In Phase I, healthy participants are not expected to benefit directly from the trial aside from the potential theoretical benefit of a mucosal immune response against SARS-CoV-2. Currently, no clinical trial data exist for a nasal protein vaccine in humans.

The anticipated risks primarily include local nasal reactions and systemic reactions similar to those observed with other vaccines. Any adverse events following vaccination are expected to be manageable with routine care, as determined by investigators.

Given that this is the first human trial of a nasal protein vaccine, the dose-escalation design ensures a safety margin, allowing for careful monitoring before progressing to the next cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the participant.
2. Be male or female between the ages of:

   1. ≥ 18 and ≤ 55 years for phase I
   2. ≥ 18 and ≤ 60 years for phase II.
3. Good general health as determined at the discretion of the investigator (vital signs, medical history, and physical examination).
4. BMI: 18,5 kg/m² ≤ BMI ˂30 kg/m².
5. Received at least 3 doses of a COVID-19 mRNA vaccine, last booster dose received at least 6 months prior to trial vaccine administration OR 2 doses of a COVID-19 mRNA vaccine and confirmed SARS-CoV-2 infection at least 6 months prior to inclusion in the trial.
6. Has expressed interest and availability to meet the trial requirements.
7. For a woman of childbearing potential, plan to be non-pregnant AND use of highly effective contraception from screening until the end of the trial.
8. Agree to abstain from donating blood/plasma or any other bodily fluids from the time of vaccination until 1 year after vaccination (only for LVT-001 vaccine).
9. Agree to stay in the geographical area of one of the clinical sites for the duration of the trial.
10. Agree to implement barrier measures as much as possible (washing hands and wearing a mask) against COVID-19 and respiratory infections between D0 and D28.
11. Agree to be registered in the computerized file of the Ministry of Health (VRB).
12. Be affiliated to French social security system.

Exclusion Criteria:

1. Temperature ≥ 38.0°C or symptoms of acute self-limiting illness such as upper respiratory tract infection or gastroenteritis within three days prior to vaccine dose.
2. Any form of contraindication to the trial vaccines tested.
3. History of chronic rhinitis, nasal septal defect, cleft palate, nasal polyps, or other nasal abnormality that might alter nasal mucosa and affect vaccine response.
4. A piercing or obstruction in the nostrils that could impede vaccine administration.
5. Previous nasal surgery or nasal cauterization.
6. History of frequent epistaxis.
7. Virologically documented (PCR or antigenic test) history of COVID-19 in the past 6 months.
8. Positive COVID-19 PCR test at screening visit.
9. Medical problems due to alcohol.
10. Illicit drug use within the past 12 months.
11. Participation in another trial within 60 days prior to the enrolment visit or planned participation during the present trial period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.

    Note: Participation in an observational study is allowed.
12. Received influenza vaccination within 14 days prior to trial vaccination, or any other licensed vaccine within 4 weeks prior to study vaccination.
13. Vaccination with a COVID-19 vaccine other than mRNA vaccine.
14. Known sensitivity to any of the ingredients of the trial vaccines.
15. Known allergic reaction to plastic.
16. Positive serology for hepatitis B (HBsAg), C (anti-HCV antibodies) and HIV 1-2.
17. History of severe adverse events following vaccine administration including anaphylactic reaction and associated symptoms such as rash, breathing problems, angioedema, and abdominal pain, or a history of allergic reaction that could be triggered by a component of the SARS-CoV-2 vaccine at the time of the first vaccine administration.
18. Pregnancy positive test (βHCG test) or pregnancy or breastfeeding.
19. Received immunoglobulin or other blood products within three months prior to inclusion or planned administration before the trial completion.
20. Received an immunosuppressive therapy for underlying disease or a treatment with immunosuppressive or cytotoxic drugs or a cancer chemotherapy or radiation therapy within the previous 36 months.
21. Received drugs such as corticosteroids at a dosage > 10 mg prednisone equivalent/day or inhalers corticosteroids, within 3 months prior to inclusion (excluding corticosteroid topical preparations for cutaneous application).
22. Abnormal and deemed clinically significant result by the investigator following the routine analyzes carried out at the time of the screening visit (any grade 4 biological result, even if deemed not clinically significant by the investigator, constitutes an exclusion criterion).
23. History of severe psychiatric disorders that may affect participation in the trial.
24. Any other serious chronic illness requiring immediate monitoring by a hospital specialist.
25. Any other condition that, in the opinion of the investigator, would compromise the safety or rights of a volunteer participating in the trial or render the subject unable to comply with the protocol.
26. Phase II only: Participants included in phase I will not be included in phase II.
27. Participants under legal protection (e.g., guardianship, tutorship).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Phase I: Proportion of participants experiencing an immediate adverse event | Within an hour and half following the vaccination at Day 0
Phase I: Proportion of participants experiencing solicited local reactogenicity | Between Day 0 and Day 7 (Day 0 is the day of the vaccination)
  Vaccines are associated with a number of well-characterised reactions referred to as "solicited adverse events"
Phase I: Proportion of participants experiencing solicited systemic signs and symptoms | Between Day 0 and Day 14 (Day 0 is the day of the vaccination)
  Vaccines are associated with a number of well-characterised reactions referred to as "solicited adverse events"
Phase I: Proportion of participants experiencing an unsolicited adverse events | Between Day 0 and Day 28 (Day 0 is the day of the vaccination)
  Unsolisited adverse events (AEs) are AEs other than solicited AEs
Phase I: Proportion of participants experiencing serious adverse events (SAEs), serious adverse reactions (SARs), suspected unexpected serious adverse reactions (SUSARs) and adverse events of special interest (AESI) respectively throughout the study | Between Day 0 to Month 12 (Day 0 is the day of the vaccination)
Phase II: Crude variation of the mucosal humoral immune response specific to the vaccine N/S recombinant protein in each arm | Between Day 0 and Day 28 (Day 0 is the day of the vaccination)
  sIgA from nose swabs measured by ELISA

SECONDARY OUTCOMES:
Crude variation of the mucosal humoral immune response specific to the vaccine N/S recombinant protein | Between Day 0 and Day 7 (Phase I), Day 14, D28 (Phase I), Month 3, Month 6 and Month 12 (Day 0 is the day of the vaccination)
  sIgA from nose swabs measured by ELISA
Neutralizing capacity of the mucosal humoral immune response specific to the vaccine N/S recombinant protein | At Day 0, Day 7 (Phase I), Day 14, Day 28, Month 3, Month 6, Month 12 (Day 0 is the day of the vaccination)
  Neutralizing Ig from nose swabs measured by PRNT and VLP assays
Crude variation of the systemic humoral immune response specific to the vaccine N/S recombinant protein | At Day 0, Day 7 (Phase I), Day 14, Day 28, Month 3, Month 6, Month 12 (Day 0 is the day of the vaccination)
  Serum anti-S and anti-N IgG measured by ELISA
Neutralizing capacity of the systemic humoral immune response specific to the vaccine N/S recombinant protein | at Day 0, Day 7 (Phase I), Day 14, Day 28, Month 3, Month 6, Month 12 (Day 0 is the day of the vaccination)
  Neutralizing serum IgG measured by PRNT and VLP assays
Percentage of responder against N and S antigens | at Day 0, Day 7 (Phase I), Day 14, Day 28, Month 3, Month 6, Month 12 (Day 0 is the day of the vaccination)
  Quantification of IFN-gamma specifically secreted by T lymphocytes following exposure to antigens N and S measured by ELISpot SARS-CoV-2 assay (subset of participants recruited only in the Tours site for feasibility reason - Phase I: 6 participants in each dose group. Phase II: 40 participants)
Proportion of participants with COVID-19 infections confirmed by a positive PCR test or a positive antigen test in each arm | Between Day 0 and Month 12 (Day 0 is the day of the vaccination)
Description of variant types identified on participants with a positive PCR test | In case of positive PCR test between the vaccination on Day 0 and Month 12
Proportion of participants with serious COVID-19 infections defined as a hospitalization and/or death due to the COVID-19 | Between Day 0 and Month 12 in each arm (Day 0 is the day of the vaccination)
Phase II: Proportion of participants experiencing an immediate AE | Within one hour following the vaccination at Day 0
Phase II: Proportion of participants experiencing solicited local reactogenicity | Between Day 0 and Day 7 (Day 0 is the day of the vaccination)
  Vaccines are associated with a number of well-characterised reactions referred to as "solicited adverse events"
Phase II: Proportion of participants experiencing solicited systemic signs and symptoms | Between Day 0 and Day 14 (Day 0 is the day of the vaccination)
  Vaccines are associated with a number of well-characterised reactions referred to as "solicited adverse events"
Phase II: Proportion of participants experiencing an unsolicited adverse events | Between Day 0 and Day 28 (Day 0 is the day of the vaccination)
  Unsolisited adverse events (AEs) are AEs other than solicited AEs
Phase II: Proportion of participants experiencing serious adverse events (SAEs), serious adverse reactions (SARs), suspected unexpected serious adverse reactions (SUSARs) and adverse events of special interest (AESI) respectively throughout the study | Between Day 0 and Month 12 (Day 0 is the day of the vaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Zoha MAAKAROUN-VERMESSE, Dr., Study Chair — University Hospital, Tours; Odile LAUNAY, Prof., Study Chair — Cochin Hospital, Paris, France; Isabelle DIMIER-POISSON, Prof., Study Chair — University, Tours, France
Locations (5):
- France (5):
  - CHU Dijon Bourgogne - Centre d'Investigation Clinique 1432, Dijon
  - HCL - Hôpital de la Croix-Rousse - Service des Maladies Infectieuses et Tropicales, Lyon
  - APHP - Hôpital Cochin - Centre d'Investigation Clinique de Vaccinologie Cochin-Pasteur 1417, Paris
  - CHU de Saint-Etienne - Service des Maladies Infectieuses, Saint-Priest-en-Jarez
  - CHRU de Tours - Centre d'Investigation Clinique 1415, Tours

IPD SHARING:
Plan to Share IPD: Undecided